CLINICAL TRIAL: NCT02769507
Title: Transcranial Brain Stimulation and Its Underlying Neural Mechanisms as a Novel Treatment for Auditory Hallucinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bergen (Other)
Collaborators: Helse-Bergen HF (Other)
Responsible Party: Principal Investigator, Marco Hirnstein, PhD, University of Bergen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UiB-BFS-01/2016
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Psychotic Disorders
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- real tDCS (Experimental): DC Stimulator PLUS (NeuroConn) The real tDCS condition comprises two daily sessions of 20 min tDCS, separated by a minimum break of 3h, for five consecutive days. Anodal and cathodal tDCS will be applied with 2mA to the left dorsolateral prefrontal cortex (a point midway between F3 and FP1) and the left peri-Sylvian region (a point midway between T3 and P3), respectively. Electrode size is 7cm x 5cm.
  Interventions: Device: DC Stimulator PLUS (NeuroConn)
- sham tDCS (Sham Comparator): DC Stimulator PLUS (NeuroConn) The sham condition is identical to the "real tDCS" condition except that after 40s of tDCS stimulation is going to be reduced to a small pulse every 550msec (110 μA over 15 msec) through the remainder of the 20 minute period.
  Interventions: Device: DC Stimulator PLUS (NeuroConn)

INTERVENTIONS:
Device: DC Stimulator PLUS (NeuroConn)

SUMMARY:
The present study aims to investigate whether transcranial direct current stimulation (tDCS) reduces auditory hallucinations in patients with psychosis. In addition, the neuronal changes of tDCS will be examined.

DETAILED DESCRIPTION:
The majority of patients with psychosis experience hallucinations, particularly auditory hallucinations are frequent. The hallucinations often leads to massive distress and impairments in social functioning and sometimes even order patients to commit acts of violence against themselves or others. The standard treatment for auditory hallucinations is antipsychotic medication. However, side-effects can be severe and about 25-30% of the patients do not respond to the medication. Transcranial direct current stimulation is a non-invasive brain stimulation technique, which modulates cortical excitability in a pain-free free with mild transient adverse effects, if any. Typically, cortical excitability underneath the anode is boosted while cathodal stimulation has inhibitory effects. Previous studies found that 2 daily sessions of 20 min tDCS for five subsequent days may reduce auditory hallucinations. Investigators want to further assess the efficacy of tDCS in sample that is large enough to detect medium to large effects. In addition, investigators want to investigate the neural mechanisms that underlie the tDCS treatment by examining various neuroimaging parameters before, immediately after treatment, and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia spectrum disorder or other psychotic disorder
* Frequent auditory hallucinations (at least 5 times a week).
* Patients are on a stable dose of antipsychotic medication (which can also be zero) for at least 2 weeks.
* Mentally competent for informed consent.
* Provided informed consent.

Exclusion Criteria:

* Metal objects in or around the head that cannot be removed (i.e. cochlear implant, surgical clips, piercing)
* History of seizures, or a history of seizures in first-degree relatives.
* History of eye trauma with a metal object or professional metal workers
* History of brain surgery, brain infarction, head trauma, cerebrovascular accident, broken skull, brain tumour, heart disease, cardiac pacemaker.
* Skin disease on the scalp on the position of the tDCS electrodes
* Coercive treatment based on a judicial ruling
* Pregnancy in female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Auditory Hallucination Rating Scale (AHRS) | Change from Baseline to immediately after treatment and 3 months after treatment
  Measure for severity of hallucinations
Questionnaire for Psychotic Experiences (QPE) | Change from Baseline to immediately after treatment and 3 months after treatment
  Measure for severity of hallucinations
Positive and Negative Syndrome Scale (PANSS) | Change from Baseline to immediately after treatment and 3 months after treatment
  Measure for positive and negative symptoms in psychotic disorders
Hallucinations App | Continuously between baseline and 3 months after treatment
  iPhone/iPod application for self-ratings of auditory hallucinations
Hallucination Change Scale (HCS) | Change from Baseline to immediately after treatment and 3 months after treatment
  Measure for changes in severity of auditory hallucinations

SECONDARY OUTCOMES:
Stroop task | Change from Baseline to immediately after treatment and 3 months after treatment
  Measure of executive functioning
Trailmaking test A and B | Change from Baseline to immediately after treatment and 3 months after treatment
  Measure of visuomotor speed
Expectations Questionnaire | Change from Baseline to immediately after treatment and 3 months after treatment
  prior expectations participants have regarding the outcome of the treatment on a scale from 0 ("The treatment will have no effect") to 10 ("The treatment will make the voices go away entirely.")
Adverse Effects Questionnaire | The questionnaire is completed after each tDCS session. That is, twice on each day of the five day treatment program
  The presence and severity of side-effects will be monitored using the tDCS adverse effects questionnaire
The Clinical Global Impressions Scale - Severity | Change from Baseline to immediately after treatment and 3 months after treatment
  Measure of global functioning
Global Assessment of Functioning | Change from Baseline to immediately after treatment and 3 months after treatment
  Measure of global functioning
Shape, size, and integrity of gray and white matter structures in the brain | Change from Baseline to immediately after treatment and 3 months after treatment
  Structural Magnetic Resonance Imaging (MRI)
GABA and glutamate levels in the dorsolateral prefrontal cortex and peri-Sylvian regions | Change from Baseline to immediately after treatment and 3 months after treatment
  MR spectroscopy
BOLD (Blood Oxygenation Level Dependent signal) response during resting state | Change from Baseline to immediately after treatment and 3 months after treatment
  Resting state functional MRI
Dichotic listening paradigm | Change from Baseline to immediately after treatment and 3 months after treatment
  Measure of executive functioning
Dichotic listening paradigm | Change from Baseline to immediately after treatment and 3 months after treatment
  Measure of language lateralization
BOLD response during dichotic listening paradigm | Change from Baseline to immediately after treatment and 3 months after treatment
  Changes in brain activity in the left dorsolateral prefrontal cortex and the peri-Sylvian language regions
White matter structure and connectivity | Change from Baseline to immediately after treatment and 3 months after treatment
  MR Diffusion Tensor Imaging

CONTACTS AND LOCATIONS:
Overall Officials: Marco Hirnstein, PhD, Principal Investigator — University of Bergen
Locations (1):
- University of Bergen, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with the ERC Advanced Projects Advanced Grant #249516 "VOICE" and #693124 "ONOFF".